CLINICAL TRIAL: NCT00002588
Title: Phase I Trial of Sequential Topotecan(NSC 609699)and Etoposide for Patients With Relapsed, Refractory,or High Risk Acute Myeloid or Lymphoid Leukemia
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Brenda W. Cooper, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2994; P30CA043703 (NIH); CWRU-ICC-2994 (Other: Case Comprehensive Cancer Center); NCI-T94-0078D
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Leukemia, Erythroblastic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Etoposide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: etoposide
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of topotecan and etoposide in treating patients who have recurrent or refractory leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of topotecan when combined with etoposide in patients with relapsed or refractory acute myelogenous leukemia, acute lymphoblastic leukemia, or blastic phase chronic myelogenous leukemia. II. Determine the toxicity of this regimen in these patients. III. Measure serum levels of topotecan at steady state and correlate them with any change in topoisomerase II content in leukemic blasts. IV. Assess whether it is feasible to correlate any upregulation of topoisomerase II expression with tumor response to etoposide in subsequent Phase II studies. V. Assess whether levels of pretreatment expression of topoisomerases I and II in leukemic cells are predictive of clinical response. VI. Assess whether it is feasible to develop a pharmacodynamic assay based on posttreatment apoptotic changes in leukemic blasts and whether this could be correlated with tumor response in subsequent phase II trials. VII. Determine the response in patients treated with this regimen.

OUTLINE: Induction: 2-Drug Combination Chemotherapy. Topotecan, TOPO, NSC-609699; Etoposide, VP-16, NSC-141540. Consolidation: 2-Drug Combination Chemotherapy. TOPO; VP-16.

PROJECTED ACCRUAL: 15-23 patients will be accrued in approximately 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myelogenous leukemia (M0-M7) and acute lymphoblastic leukemia (L1-L2) Refractory or in first or subsequent relapse Circulating blasts present OR Greater than 5% blasts in bone marrow Acute myelogenous leukemia secondary to myelodysplastic syndrome or cytotoxic therapy Untreated OR Maximum of 2 intensive induction regimens Chronic myelogenous leukemia in blastic or lymphoid crisis Untreated OR Maximum of 2 intensive induction regimens No CNS leukemia

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-3 Life expectancy: At least 4 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL AST and ALT less than 3 times normal Alkaline phosphatase less than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No myocardial infarction within 6 months No active ischemic cardiac disease No poorly controlled congestive heart failure No other symptomatic cardiac disease Left ventricular ejection fraction at least 40% Pulmonary: No symptomatic restrictive or obstructive lung disease Other: No severe neurologic disease No active infection unless stable on antimicrobial therapy or fever is tumor related HIV negative Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: At least 2 weeks since prior cytotoxic therapy (except hydroxyurea and steroids) Biologic therapy: No prior bone marrow transplantation At least 3 days since prior hematopoietic growth factors Chemotherapy: No prior topotecan or camptothecin analogues Prior etoposide allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1994-08; Primary Completion 2000-07 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of topotecan when combined with etoposide in patients with relapsed or refractory acute myelogenous leukemia, acute lymphoblastic leukemia, or blastic phase chronic myelogenous leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda W. Cooper, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Cooper BW, Lazarus HM, Creger R, et al.: A phase I and pharmacodynamic study of sequential topotecan and etoposide (TE) in adult patients with refractory/relapsed acute leukemia (RAL) (Meeting abstact.). [Abstract] Proceedings of the American Society of Clinical Oncology 15: A1549, 1996.